CLINICAL TRIAL: NCT07030192
Title: Promoting Safety and Equity in Chaos: A Feasibility Study of Peer Support Workers to Support People Who Use Drugs in Emergency Departments
Brief Title: Peer Support Workers Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Coastal Health Research Institute (Other); BC Centers for Disease Control (Unknown)
Responsible Party: Principal Investigator, Jessica Moe, Assistant Professor UBC Department of Emergency Medicine, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H24-03008
Record Dates: First submitted 2025-06-03; First posted 2025-06-22 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Substance Use Disorder (SUD)
Keywords: Peer support workers; Substance use; Emergency department
MeSH Terms: conditions — Substance-Related Disorders; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer support service (Experimental): Patients presenting with substance use related complaints during days and times where a Peer is available to provide services, as per an a priori, randomized schedule
  Interventions: Behavioral: Peer support service
- No Peer intervention (No Intervention): Patients with substance use presentations who present to EDs on days and times when a Peer is not available, as per an a priori, randomized schedule

INTERVENTIONS:
Behavioral: Peer support service — Peers approach identified patients who could potentially benefit from peer support services. Peers offer a range of supports tailored to individual patients' needs, which include referrals to clinical and social support services (e.g., social work, addictions specialist, Indigenous patient navigator, community-based addictions resources), resources (e.g., blankets, food, naloxone kit, sterile drug use supplies, information brochures), providing emotional support, and liaising between patients and healthcare providers to communicate information about patients' condition and ED trajectory.
  Peer support workers share their personal experiences to guide patients through their ED visit and to facilitate awareness and understanding of available resources.
  Arms: Peer support service

SUMMARY:
Many people with high-risk opioid use visit emergency departments (EDs), facing a high risk of death if they leave before completing care. Peer support workers (Peer) - people with lived experience of substance use - may improve patient comfort, reduce early departures, and potentially lower mortality rates. This study aims to evaluate how a hospital-implemented ED Peer program can enhance patient support, reduce barriers to care, and provide harm-reduction resources in a person-centred and trauma-informed manner. The study will also validate the outcome and obtain preliminary estimates of the benefits of decreasing patients who leave the ED before completing care.

DETAILED DESCRIPTION:
The main objectives of the study are to 1) to describe, and evaluate the feasibility and acceptability of a novel ED Peer program implemented by the Vancouver Coastal Health at the Vancouver General Hospital (VGH) ED, 2) to evaluate the feasibility of creating a randomized shift schedule in support of a future definitive randomized controlled trial, 3) to validate outcomes related to patients leaving before completing care using administrative data from the National Ambulatory Care Reporting System (NACRS), and 4) to obtain preliminary estimates of incidence of patients who leave the ED before completing care, to inform sample size calculations for a definitive randomized controlled trial.

The study will take place at Vancouver General Hospital (VGH), a large ED with approximately 97,000 visits per year, serving a diverse urban population. Investigators will evaluate our randomized shift schedule generation, and will describe our intervention and patient population through data within our Peer interaction logs and linkages to regional data. To understand our intervention and patient and provider experiences, investigators will use a mixed methods design to comprehensively collect, analyze, and interpret both qualitative and quantitative data. This approach will provide insights from multiple perspectives, offering a robust understanding of the relationships and potential contradictions within the evidence, thereby enriching the data and deepening our understanding of the findings.

Investigators will evaluate feasibility and acceptability of the Peer program at engaging patients with specific demographic, health history, and risk profiles. Investigators will assess the degree to which patients of different backgrounds access and engage with Peer services, and what characteristics affect patient acceptance of Peer services offered. Investigators will then work with the ED leadership team to target and tailor the program to best meet the needs of patients at highest risk.

This feasibility study will set the foundation for a definitive randomized controlled trial, which will be the first to compare patients with substance use who leave EDs before completing care during shifts with Peer availability versus without, addressing a critical knowledge gap. The definitive trial will engage multiple sites across Canada to rigorously evaluate ED Peer effectiveness, with the potential to scale up an intervention that could improve patient outcomes on a national scale.

ELIGIBILITY:
Inclusion Criteria:

* Emergency Department (ED) patient at Vancouver General Hospital (VGH)
* Age 18 years or older
* Identified as using substances
* Able to receive or decline peer support services during the ED visit

Exclusion Criteria:

* Under 18 years of age
* Does not report substance use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3181 (Estimated)
Dates: Start 2024-11-23 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Distribution of randomized Peer shifts by day of week | Over the 48-week randomized schedule period approved to meet hospital staffing policy
  Assessed by examining the distribution of scheduled Peer shifts across each day of the week over the 48-week randomized schedule period. The schedule was developed in collaboration with human resources and ED operational leadership and approved as meeting hospital employee policy. The randomization approach used block-based scheduling with built-in constraints (e.g., mandatory weekends off). This outcome evaluates whether the resulting schedule achieved an even weekday/weekend distribution.
  Unit of Measure: Number and percentage of Peer shifts scheduled per day of the week
Proportion of Peer interactions with complete standardized documentation | Up to 15 months post-study initiation
  Assessed by the proportion of Peer interactions that were fully recorded using the standardized Peer interaction log, with completion defined by filling all required fields.
  Unit of Measure: Percentage of interactions with complete logs
Identification of substance use-related ED visits for Peer and No Peer shift comparison | Up to 15 months post-study initiation
  Investigators will obtain regional ED data with all visit information on all ED visits made during our study period. Investigators will use randomized schedule to identify dates and times of Peer shifts and control shifts. Investigators will then assess proportion of patients who left before medically advised among those presenting with substance use-related complaints during times with ED Peers available, compared to times without Peers. Investigators will analyze patients with presenting complaints that denote common complications of substance use (localized swelling/redness, substance withdrawal, and substance misuse/intoxication). This cohort can be identified using administrative data alone, allowing investigators to identify a reliable comparator group when ED Peers are not present. .
Characterization of Patients Receiving the Peer Intervention | Baseline. Up to 15 months post-study initiation.
  Investigators will describe characteristics of patients who received the Peer intervention using information from interaction logs (including sex and gender) and linked administrative data (e.g., preceding substance use-related encounters; databases described below).
Patients leaving the ED prior to completing care | Baseline. Data will be linked and assessed at the conclusion of the feasibility study, up to 15 months post-study initiation.
  Investigators will use a linear regression model to compare the shift-level percentage of visits resulting in left before medically advised(primary outcome) during intervention (Peer) and control (no Peer) shifts, among all visits made by patients with our presenting complaints of interest. Patients presenting in the Peer shifts will be included in the analysis irrespective of whether they received the Peer intervention, i.e., an intent-to-treat approach. The model will adjust for shift-level covariates including: day of week, shift type (morning/afternoon/night), and ED volume.
"Treatment effect in the treated" analysis | Up to 15 months post-study initiation
  Investigators note that the shift-level analysis includes many patients who are not targets for the intervention. This is unavoidable because the absence of screening in the control arm renders it impossible to identify who would be eligible for the intervention, but including non-target patients introduces noise into the analysis and dilutes the observed effect. Hence, investigators will use a mixed-effect logistic regression at the patient level to compare the probability of left before medical advice in patients who presented with a specific complaint (e.g., substance misuse) and received the intervention, to patients in the control arm who presented with the same complaint. Investigators will use medical record numbers collected by Peers as part of the interaction logs to identify people who interacted with a Peer. The model will adjust for age, sex, time of day, day of week, month, ambulance arrival, triage acuity, and presenting complaint.

SECONDARY OUTCOMES:
Thematic summary of Indigenous patients' experiences with the Peer program based on storytelling and sharing circles | Within 6 months after the patient's ED visit involving Peer interaction
  Indigenous patient perspectives on the Peer program will be collected through culturally grounded storytelling and sharing circles. Sessions will be guided by open-ended questions to explore perceived safety, support, and emotional impact of Peer involvement in the emergency department. Transcripts will be analyzed using Indigenous-informed thematic analysis to identify key insights and priorities for culturally safe care.
  Unit of Measure: Themes and narratives identified through qualitative analysis
Thematic summary of healthcare providers' perceptions of the Peer program assessed through focus groups | From 3 to 15 months after program implementation
  Acceptability of the Peer program among healthcare providers will be evaluated using semi-structured focus groups conducted between 3-15 months post-implementation. Discussions will explore perceived value, observed patient impact, integration into ED workflows, challenges, and suggestions for improvement. Audio recordings will be transcribed and analyzed using thematic content analysis to identify recurring patterns and representative quotes.
  Unit of Measure: Thematic categories identified through qualitative analysis
Patient-reported acceptability of the Peer program using the Peer patient survey | Up to 15 months post-study initiation
  Acceptability will be assessed using the Peer patient survey, a 15-item questionnaire completed by patients following interaction with a peer support worker. Each item is scored on a 5-point Likert scale ranging from 1 (Strongly Disagree) to 5 (Strongly Agree). Items assess patient experiences related to respect, emotional safety, ease of communication, clarity of information, comfort, confidentiality, and teamwork. The primary reported outcome will be the mean overall score across all 15 items. Secondary analyses may report item-level distributions.
  Unit of Measure: Mean overall score (1-5 scale).
  Scale Range: 1 (Strongly Disagree) to 5 (Strongly Agree); higher scores indicate higher acceptability of the Peer program.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Moe, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers